CLINICAL TRIAL: NCT07026721
Title: Comparative Analysis of RIRS Scoring System and Resorlu Unsal Stone Score (RUSS) for Predicting Stone-Free Rate After Retrograde Intrarenal Surgery: A Prospective Cohort Study
Brief Title: Comparative Analysis of RIRS Scoring System and Resorlu Unsal Stone Score (RUSS) for Predicting Stone-free Rate After Retrograde Intrarenal Surgery
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Prajjwol Luitel, Principal Investigator, Maharajgunj Medical Campus
Other Study IDs: 407(6-11)E2.080.081
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-01

CONDITIONS: Renal Stones
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery (RIRS) — The intervention involves Retrograde Intrarenal Surgery (RIRS) performed using a flexible ureteroscope to access the renal collecting system via a retrograde (urethra → bladder → ureter → kidney) approach. Stones are fragmented using a holmium:YAG laser, with or without the use of a ureteral access sheath, depending on the case.
  What distinguishes this intervention from others is the integration of preoperative scoring systems-specifically the RIRS Scoring System and the Resorlu Unsal Stone Score (RUSS)-to predict stone-free outcomes and guide case selection and surgical planning. Additionally, all procedures are performed by experienced endourologists following a standardized protocol, including consistent patient positioning, anesthesia, access technique, and post-operative imaging at defined intervals to assess outcomes.

SUMMARY:
Several studies have investigated the use of scoring systems for predicting stone-free rates after RIRS. Previous research has evaluated the RIRS Scoring System, RUSS, and other similar systems in different patient populations. This study was conducted to compare RIRS scoring system and Resorlu Unsal Stone Score (RUSS) for predicting stone free rate.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years of age undergoing RIRS for renal stone
* providing informed written consent

Exclusion Criteria:

* Previous renal and ureteric surgeries
* coexisting bladder, ureteral stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with renal calculi undergoing RIRS.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Correlation between the RIRS Scoring System and stone-free rate after Retrograde Intrarenal Surgery (RIRS), assessed using CT KUB | 12 months
Correlation between the Resorlu-Unsal Stone Score (RUSS) and stone-free rate after Retrograde Intrarenal Surgery (RIRS), assessed using CT KUB | 12 months

SECONDARY OUTCOMES:
Stone Burden as a Predictor of Stone-Free Rate After RIRS | Preoperative assessment and 1 month postoperatively for stone-free status
  Correlation between stone burden (mm²) and stone-free rate after Retrograde Intrarenal Surgery (RIRS
Stone Density as a Predictor of Stone-Free Rate After RIRS | Preoperative assessment and 1 month postoperatively for stone-free status
  Correlation between stone density (Hounsfield Units, HU) and stone-free rate after RIRS

CONTACTS AND LOCATIONS:
Overall Officials: Saro Prajapati, MBBS, MS, Study Director — Department of General Surgery Maharajgunj Medical Campus Institute of Medicine, Tribhuvan University
Locations (1):
- Department of Urology and Kidney Transplant Surgery, Tribhuvan University Teaching Hospital (TUTH), Maharajgunj, Kathmandu, Nepal, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol